CLINICAL TRIAL: NCT03323879
Title: Dominant Intraprostatic Lesion Boost With Focused LDR Brachytherapy (BT) Integrated to Whole Prostate HDR BT: Safety and Feasibility Analysis
Brief Title: Combined LDR Boost and HDR Whole Gland
Acronym: Delight
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DELIGHT
Record Dates: First submitted 2017-09-12; First posted 2017-10-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma Prostate
Keywords: brachytherapy; LDR; HDR; monotherapy; focal
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDR/HDR (Experimental): MRI planned LDR boost to DIL with concurrent whole gland 19 Gy HDR. LDR dose will be sequentially escalated from 50 Gy to 80 Gy
  Interventions: Radiation: LDR/HDR

INTERVENTIONS:
Radiation: LDR/HDR — Focal LDR to dominant lesion with whole gland 19 Gy HDR

SUMMARY:
This is a dose finding Phase I/II study of combined focused LDR brachytherapy boost with whole gland single fraction HDR for men with low and intermediate risk prostate cancer and Dominant Intraprostatic Lesion (DIL) visible on multi parametric MRI. Patients will receive 19 Gy HDR to the whole gland with concurrent LDR brachytherapy boost to the DIL, in a sequential dose escalation manner. Primary endpoints are early toxicity.

DETAILED DESCRIPTION:
Eligible patients will have low and intermediate risk prostate cancer with a dominant intraprostatic lesion definable on multi parametric MRI (PIRADS 4 or 5). Patients will have MR planned LDR focal brachytherapy to the DIL using iodine-125, while at the same time have single 19 Gy delivered to the whole prostate using ultrasound directed high dose-rate brachytherapy (HDR). The LDR boost dose will start at 50 Gy, and increase DIL dose in sequential cohorts of patients up until a dose of 80 Gy. Up to 20 patients will be included. Primary endpoint is toxicity at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Adenocarcinoma of the prostate
* Single PIRADS 4 or 5 lesion on multiparametric MRI
* T1c-T2b on rectal exam
* Gleason 3+3 and PSA < 20ng/mL
* Gleason 3+4 and PSA <10ng/mL
* Less than 50% of the cores positive in an untargeted prostate biopsy.
* Prostate volume < 60 cc

Exclusion Criteria:

* Incapable or ineligible for MRI imaging
* Previous trans-urethral resection of prostate (TURP)
* Previous or current use of androgen deprivation
* Baseline International Prostate Symptom Score (IPSS) > 15
* Evidence of distant or nodal metastasis
* Disease that contraindicates treatment with radiation (e.g connective tissue disease)
* Unsuitable for anesthesia due to comorbidity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Acute urinary and rectal toxicity at 3 months as measured using NCI CTCAE v 4.0 | At 3 months
  Acute urinary and rectal toxicity within the first 3 months as measured using NCI CTCAE v4.0

SECONDARY OUTCOMES:
Late urinary and rectal toxicity using NCI CTCAE v4.0 | 3-monthly for first year, then 6-monthly until Year 5
  Cumulative incidence of urinary and rectal toxicity beyond 3 months using NCI CTCAE v4.0.
Health related quality of life (HRQOL) changes | 3 monthly for first year, then annually year 1-5
  Changes in HRQOL as assessed using Expanded Prostate Index Composite (EPIC)
Disease Free Survival | will be reported at 5 years
  biochemical disease-free survival using PSA nadir + 2 ng/ml definition (Phoenix)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided